CLINICAL TRIAL: NCT02341248
Title: Gut Microbial Taxonomy and Metabolism in Paediatric Crohn's Disease During Exclusive and Supplementary Enteral Nutrition Using -Omics Technologies
Brief Title: Bacteria & Inflammation in the Gut (BIG) Study
Acronym: BIG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: GN14KH275
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Crohn Disease
Keywords: Enteral Nutrition; Pediatrics; Microbiota; Metabolomics
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, faecal, urine and mucosal samples retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A) Newly diagnosed with Crohn's disease: Children undergoing endoscopic investigations (colonoscopy) for colonic inflammation including Crohn's disease [children who are found not to have Crohn's disease will not participate further].
  [Intervention - clinical, not research decision - Exclusive Enteral Nutrition for 8 weeks; usually 330ml 6 times per day] per day
  Interventions: Other: Exclusive Enteral Nutrition (EEN)
- B) Existing diagnosis of Crohn's disease: Previously diagnosed patients with Crohn's disease due to start an 8 week standard course of treatment with EEN due to disease flare up.
  [Intervention - clinical, not research decision - Exclusive Enteral Nutrition for 8 weeks; usually 330ml 6 times per day]
  Interventions: Other: Exclusive Enteral Nutrition (EEN)
- c) Healthy control group: Healthy children unrelated to Crohn's disease patients No intervention

INTERVENTIONS:
Other: Exclusive Enteral Nutrition (EEN) — 8 week standard course of treatment with EEN
  Groups: A) Newly diagnosed with Crohn's disease; B) Existing diagnosis of Crohn's disease

SUMMARY:
Exclusive Enteral Nutrition (EEN) is the liquid diet given to children with active Crohn's Disease (CD). EEN has previously been shown to induce changes in major bacterial metabolites and dominant bacterial species which are more profound in children that clinically improve. This study aims to determine whether it is possible to maintain these bacterial changes with prolonged supplementary enteral nutrition (SEN) while returning to normal diet and if this can reduce risk of subsequent relapse for children with CD.

New technologies will allow measurement of a broad range of bacteria and metabolites, to test if the clinical response to EEN and changes in gut inflammation are associated with bacterial composition and chemical products; and if maintenance of changes using SEN reduces the risk of relapse over a 12 month period.

The study will aim to recruit all potential Crohn's disease children coming to a tertiary paediatric centre for colonoscopy. Once consented, an initial blood, urine and faecal sample will be requested along with 8 mucosal biopsies during the routine endoscopy session. If diagnosed with CD, and if the clinician prescribes treatment with EEN, an additional blood sample will be requested at the end of EEN, and 5 faecal and urine samples spread over 12 months; as well as some dietary information.

Samples will be collected from up to 42 children with CD and 42 age- and sex-matched healthy volunteers. Initial samples taken from children who were not diagnosed with CD will be compared with CD samples to look for potential metabolic disease markers. Characterisation of faecal bacteria and metabolites in both faeces and urine; as well as measurement of blood inflammatory biomarkers will be performed.

DETAILED DESCRIPTION:
The null hypothesis is that the clinical response to exclusive enteral nutrition (EEN) and reduction of colonic inflammatory markers are not associated with a characteristic bacterial taxonomy (composition) and metabolites (functionality); and that maintenance of any bacterial changes with supplementary enteral nutrition (SEN), while returning to habitual diet, does not reduce the risk of disease relapse.

The study design will build on previous work by looking at differences in both the gut bacteria (faecal and mucosal) and bacterial metabolic activity at different stages of disease activity. Changes in bacterial composition between disease groups will be examined; between Crohn's disease children on different treatments; and between different sites in the gut. Crohn's disease biomarkers in faeces and urine will also be assessed by analysing bacterial metabolites.

Up to a total of 42 children with Crohn's Disease will be recruited. 42 healthy children will also be recruited to provide a faecal and urine sample, to show the normal variety of gut bacteria and metabolites in healthy children for comparison.

Children who underwent colonoscopy but did not have Crohn's disease will be used as a comparison group to try and identify Crohn's disease bacterial signatures from faeces and urine, and as a non-Crohn's disease control group for comparison of mucosal biopsies.

Recruitment Three groups of children will participate in this study. A. Children undergoing endoscopic investigations (colonoscopy) for colonic inflammation including Crohn's disease [children who are found not to have Crohn's disease will not participate in the follow up aspect (during treatment with EEN) of this study].

B. Previously diagnosed patients with Crohn's disease due to start an 8 week standard course of treatment with EEN due to disease flare up.

C. Healthy children unrelated to Crohn's disease patients will be used as a control group.

Groups A and B: an initial blood, urine, faecal sample followed by 5 further faecal and urine samples over 12 months; and dietary information.

[Group A will also have 8 mucosal biopsies taken during routine endoscopy]. During treatment with EEN (clinical decision), an additional blood sample will be requested during routine blood sampling at start and end of treatment.

Group C: 1 urine and faecal sample will be requested.

All groups will have height, weight and grip strength measured at baseline. Participant receiving EEN will have this repeated 60 days after start of treatment and 60 days after end of treatment.

Detailed Methods Preliminary health check by means of a short health questionnaire - basic health information, age, any medication.

Mucosal samples: in newly diagnosed patients having a colonoscopy for diagnostic purposes, an additional 6 mucosal biopsy samples; 2 from the terminal ileum when possible, 2 from the proximal colon and 2 from the distal colon will be taken (14-16 are collected at normal colonoscopy). An additional 2 biopsy samples will also be collected from the duodenum during upper endoscopy.

Dietary information: habitual dietary intake and eating patterns assessed using validated Food Frequency Questionnaire (FFQ); a 5 step multiple pass 24 hour dietary recall questionnaire for data on actual diet at time of faecal and urine sampling.

EEN compliance (groups A&B only): completion of short EEN compliance questionnaire at 28 day and 56 day time points.

Medication and Disease History: information on disease activity, medication and medical history collected from medical notes.

Lab Assays Bacterial diversity: The gut bacterial diversity and composition from stool samples will be measured using molecular techniques such as quantitative polymerase chain reaction (PCR) from bacterial ribosomal DNA and next generation sequencing (metagenomics). These techniques will also be used to look at the composition of bacteria associated with mucosal tissue biopsies. Changes in overall gut bacteria composition using standard numerical indices will be measured across the 6 faecal samples collected over the 12 month period, as well as between groups.

Bacterial metabolism: A large number of different products from bacterial metabolism, such as short chain fatty acids, sulphide, and ammonia will be measured using a range of techniques including gas chromatography and gas chromatography mass spectrometry (GCMS) (metabolomics). Faecal pH, a marker of bacterial fermentation, will also be measured.

Disease markers: Other disease markers and metabolites such as faecal calprotectin, will be measured from faecal samples .

ELIGIBILITY:
Inclusion Criteria:

* Group A: children with suspected Crohn's Disease with scheduled colonoscopy
* Group B: children with existing Crohn's Disease about to undergo treatment with EEN
* Group C: healthy volunteers up to age 17 years willing to provide one urine and stool sample

Exclusion Criteria:

* children who have taken antibiotics in the previous 4 weeks
* children found not to have Crohn's Disease after colonoscopy will not be required to take any further part in the study

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with suspected or diagnosed Crohn's Disease attending a tertiary paediatric centre for treatment with exclusive enteral nutrition
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-07-18 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Bacterial metabolism | 12 months
  Change in short chain fatty acid level following treatment with enteral nutrition
Gut bacterial composition | 12 months
  Change in overall gut bacteria composition following treatment with enteral nutrition
Mucosal bacterial composition | 12 months
  Change in overall bacteria composition in mucosal tissue biopsies

SECONDARY OUTCOMES:
Inflammatory markers | 12 months
  Change in faecal calprotectin level before and after treatment with EEN
Dietary information | 12 months
  Comparison of dietary composition between groups

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - NHS Greater Glasgow & Clyde - Royal Hospital for Sick Children, Glasgow
  - NHS Ayrshire & Arran - University Hospital Crosshouse, Kilmarnock
  - NHS Forth Valley - Forth Valley Royal Hospital, Larbert
  - NHS Greater Glasgow & Clyde - Royal Alexandra Hospital, Paisley
  - NHS Lanarkshire - Wishaw General Hospital, Wishaw

REFERENCES:
- [Derived] Logan M, MacKinder M, Clark CM, Kountouri A, Jere M, Ijaz UZ, Hansen R, McGrogan P, Russell RK, Gerasimidis K. Intestinal fatty acid binding protein is a disease biomarker in paediatric coeliac disease and Crohn's disease. BMC Gastroenterol. 2022 May 23;22(1):260. doi: 10.1186/s12876-022-02334-6. PMID 35606704
- [Derived] Gkikas K, Logan M, Nichols B, Ijaz UZ, Clark CM, Svolos V, Gervais L, Duncan H, Garrick V, Curtis L, Buchanan E, Cardigan T, Armstrong L, Delahunty C, Flynn DM, Barclay AR, Tayler R, Milling S, Hansen R, Russell RK, Gerasimidis K. Dietary triggers of gut inflammation following exclusive enteral nutrition in children with Crohn's disease: a pilot study. BMC Gastroenterol. 2021 Dec 3;21(1):454. doi: 10.1186/s12876-021-02029-4. PMID 34861829